CLINICAL TRIAL: NCT03853434
Title: Efficacy of Angiographic Embolization vs Non-embolization of Moderate/Poor Vascularized Vertebral Metastases on Intraoperative Bleeding During Surgery Decompression and Vertebral Stabilization. Randomized Controlled Observer- Blinded
Brief Title: Efficacy of Angiographic Embolization vs Non-embolization of Moderate/Poor Vascularized Vertebral Metastases on Intraoperative Bleeding During Surgery Decompression and Vertebral Stabilization.
Acronym: Embart
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Embart
Record Dates: First submitted 2019-01-15; First posted 2019-02-25 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Spine Metastasis; Early Goal Directed Therapy; Embolization, Therapeutic; Blood Loss
Keywords: embolization; blood loss; Early Goal Directed Therapy; spine metastasis
MeSH Terms: conditions — Hemorrhage | interventions — Embolization, Therapeutic

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Embolization (Experimental): After angiography all metastases with poor/moderate vascularization will be embolized with acrylic glue in the treatment group.
  Interventions: Procedure: Embolization
- No embolization (No Intervention): After angiography all metastasis with poor/moderate vascularization will not be embolized with acrylic glue in the control group

INTERVENTIONS:
Procedure: Embolization — Angiographic embolization
  Arms: Embolization

SUMMARY:
Although angiographic embolization has been introduced for preoperative management of spine metastases in 1975 and is suggested today by many authors in the management of such pathologies, it needs to be confirmed by RCT. It is a minimally invasive procedure, not free from complications. The recent meta-analyzes, due to the limited number of patients included are not exhaustive about the effectiveness of embolization in the reduction of the intraoperative bleeding, especially in the context of poor / moderate metastasis vascularization. We want to evaluate the efficacy of preoperative angiographic embolization of intermediate / poor vascularized spine metastases in reducing intraoperative blood loss during excision surgery.

ELIGIBILITY:
Inclusion Criteria:

* Male, Female aged 18 years and 75 years
* prognosis >6 months (Tokuhashi score ≤ 11)
* patients with lesions with moderate vascularization (grade 2)
* time between embolization and intervention >/= 48-72 h

Exclusion Criteria:

* congenital and iatrogenic hemocoagulative disorders (PT INR> 1.5, aPTT ratio> 1.25 with documented coagulation factor deficiency, PLT < 80,000 / microL or known coagulation pathologies);
* renal failure (creatinine ≥ 1.2);
* MDC iodized allergy;
* pregnancy / lactation;
* chronic ischemic heart disease;
* precluded arterial access by angiography;
* indication to emergency surgery;
* time between embolization and surgery> 72 h;
* refusal by the patient.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2028-11-30 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Intraoperative blood loss | during procedure
  volume (ml) of intraoperative blood loss volume aspirated from operative field (ml) + differential weight gauze at the end of surgery - dry gauze weight with 1g blood conversion = 0.948ml

SECONDARY OUTCOMES:
Concentration of Hemoglobin pre / post-operative | 24 hours
volume of transfused blood (ml) | intraoperatively
Correlation between primary tumor and vascularization | during angiographic procedure
correlation between the type of primary tumor and blood losses | 24 hours
technical evaluation of the final result of embolization (total - 100%, subtotal 90-80% and partial 70-50%) in relation to blood losses | during angiographic procedure
evaluation of operative time, from incision to end of suture | during procedure
incidence of complications related to transfusions; | during hospitalization
duration of the hospitalization in ICU | during hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Giancarlo Facchini, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided